CLINICAL TRIAL: NCT03196206
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of BMS- 986177 in Participants With Normal Renal Function and Participants With Moderate and Severe Renal Impairment
Brief Title: Evaluate Pharmacokinetics and Safety of BMS-986177 in Participants With Normal Renal Function and With Moderate or Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CV010-018
Record Dates: First submitted 2017-06-21; First posted 2017-06-22 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Normal Renal Function
  Interventions: Drug: BMS-986177
- Group B (Experimental): Moderate Renal Impairment
  Interventions: Drug: BMS-986177
- Group C (Experimental): Severe Renal Impairment
  Interventions: Drug: BMS-986177

INTERVENTIONS:
Drug: BMS-986177 — Oral Suspension

SUMMARY:
Assess the pharmacokinetics, safety, and tolerability of a single dose of BMS-986177 in participants with normal renal function and moderate to severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participants in Groups B and C will be classified by renal function by eGRF at screening and confirmed on Day -1
* Participants in Group A will be healthy participants as determined by no significant deviations in normal medical and surgical history and assessments
* Participants in Group A must have a body mass index of 18.0 to 32.0 kg/m2, inclusive
* Females must be of non-childbearing potential

Exclusion Criteria:

* Participants in Groups B and C cannot have an indwelling catheter for hemodialysis
* Participants in Groups B and C cannot have had, nor be waiting for, an organ transplant

Other protocol defined inclusion and exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-03-04 (Actual); Study Completion 2018-03-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 5 days
  Measured by plasma concentration
AUC from time zero to time of last quantifiable concentration (AUC (0-T)) | Up to 5 days
  Summary measures of PK parameters
AUC from time zero extrapolated to infinite time (AUC (INF)) | Up to 5 days
  Summary measures of PK parameters

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 5 days
  Safety and tolerability as measured by incidence of AEs
Incidence of Serious Adverse Events ( SAEs) | Up to 30 days
  Safety and tolerability as measured by incidence of SAEs
Change from baseline in electrocardiogram findings | Up to 5 days
  Measured by investigator assessment
Change from baseline in physical examination findings | Up to 5 days
  Measured by investigator assessment
Change from baseline in clinical laboratory test findings | Up to 5 days
  Measured by investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Clinical Pharmacology Of Miami Inc., Miami, Florida
  - Clinical Pharmacology of Miami LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- [Derived] Perera V, Abelian G, Li D, Wang Z, Zhang L, Lubin S, Bello A, Murthy B. Single-Dose Pharmacokinetics of Milvexian in Participants with Normal Renal Function and Participants with Moderate or Severe Renal Impairment. Clin Pharmacokinet. 2022 Oct;61(10):1405-1416. doi: 10.1007/s40262-022-01150-1. Epub 2022 Jul 30. PMID 35906349
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html